CLINICAL TRIAL: NCT05080062
Title: Requirements and Functional Schedule- An Intervention to Use in Painrehabilitation, to Strengthen the Collaboration Between the Healthcare, Employers and Employees
Brief Title: Requirements and Functional Schedule as a Part of Painrehabilitation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Katarina Danielsson, Chief physician, principal investigator, Uppsala University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019/01755
Record Dates: First submitted 2019-07-16; First posted 2021-10-15 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: 50 patients who are in painrehabilitation will also receive the intervention. The control Group will be based on patients from 2017 and 2018 who has underwent rehabilitation. This data will be extracted from the National register of pain rehabilitation in Sweden.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Painrehabilitation + Demand and ability protocol (Experimental): Will receive pain-rehabilitation and the intervention ( an interview called Requirements and functional Schedule, with the patients employer and an occupational therapist)
  Interventions: Behavioral: Requirements and functional Schedule
- Painrehabilitation (Active Comparator): Will receive pain-rehabilitation
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: Requirements and functional Schedule — An interview with the employee and the employer where the occupational worker is leading the interview and a pain rehabilitation-program
  Arms: Painrehabilitation + Demand and ability protocol
Behavioral: No intervention — a pain rehabilitation-program
  Arms: Painrehabilitation

SUMMARY:
Requirements and functional Schedule also calen Demand Ability Protocol (DAP) is an intervention that has been tested and found useful in occupational health service. The intervention aims to strengthen the collaboration between Health care, employers and employee. The intervention is based on a structured interview about the employers demands at work. This intervention (DAP) will in the present study be evaluated in pain rehabilitation both qualitatively and quantitatively.

DETAILED DESCRIPTION:
Description of the intervention: Demand and Ability Protocol Demand and Ability Protocol (DAP) is an intervention linked to the International Classification of Functioning, Disability and Health, and is based on the Dutch Functional Ability List and knowledge about disability in working life (Brouwer et al, 2002). The intervention has been further developed and modified in Norway and is primarily used in occupational health care services for collaboration between an employee and his or her immediate manager (Engbers & Furuland, 2006).

The intervention consists of a structured conversation between the patient and his immediate manager under the guidance of licensed medical staff (in this case REKO) with knowledge of the requirements of the patient's work and his/her current functional ability. The intervention takes about 90 minutes excluding preparation time for REKO.

DAP consider the following domains; 1) mental and cognitive ability, 2) basic skills and social ability, 3) tolerance for physical conditions, 4) ability to work dynamically, 5) ability to work statically and 6) to be able to work certain times.

Based on the above domains, a structured review is made of the balance between requirements and function in current work in order to identify possible adaptations and measures at the workplace. During the intervention, the work requirements and the patient's function/ability are identified on a three-point scale and in domains where the rating of requirements and function/ability does not match, there is thus an imbalance, and here adjustments or changed tasks may be relevant to consider increasing work ability and reducing sick leave. The intervention concludes with a summary of the situation and joint development of appropriate measures/adaptations to promote the patient's RTW. This is documented on a form, which is signed by both the patient and the manage

ELIGIBILITY:
Inclusion Criteria:

Chronic pain, has an employment

Exclusion Criteria:

no longer than 6 month of total sick-leave

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Absence from work (sickleave) measured with a question to the participants | Changes from baseline in absence from work to the end of the rehab program (average 4month)
  Less absence from work
Absence from work (sickleave) measured with a question to the participants | Changes from baseline in absence from work through study completion (average 1,5 years)
  Less absence from work

SECONDARY OUTCOMES:
Changes in EuroQol 5-dimensions questionnaire (EQ-5D) | Change from baseline in EuroQol 5-dimensions through study completion (average 1,5 years)
  Changes in quality of Life measured with the EuroQol 5-dimensions. Each combination of values has an idex value where 1 is the best quality of life. The questionnaire also includes a visual analog scale (VAS), which records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher qulaity of life
  .
Changes in EuroQol 5-dimensions | Change from baseline in EuroQol 5-dimensions to the end of the rehab program (average foru month)
  Changes in quality of Life measured with the EuroQol 5-dimensions. Each combination of values has an idex value where 1 is the best quality of life. The questionnaire also includes a visual analog scale (VAS), which records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher qulaity of life
Changes in Anxiety and depression | Change from baseline in anxiety and depression through study completion (average 1,5 years)hs)
  Changes in Hospital Anxiety and Depression Scale (HADS). The scale icludes two subscales one focusing on anxiety symptoms and one on depressive symptoms. The minimum value is 0 and the maximum value is 21 for each subscale. Higher scores means worse outcome.
Changes in Anxiety and depression | Change from baseline in anxiety and depression to the end of the rehab program (average four month)
  Changes in Hospital Anxiety and Depression Scale (HADS). The scale icludes two subscales one focusing on anxiety symptoms and one on depressive symptoms. The minimum value is 0 and the maximum value is 21 for each subscale. Higher scores means worse outcome.
Changes in sleep | Change from baseline in Insomnia Severity Index to the end of the rehab program (average four month)
  Changes in Insomnia measured with Insomnia Severity Index (ISI). The minimum value is 0 and the maximum value is 28. Higher scores indicates a worse outcome.
Changes in sleep | Change from baseline in Insomnia Severity Index through study completion (average 1,5 years)
  Changes in sleep measured with Insomnia Severity Index (ISI). The minimum value is 0 and the maximum value is 28. Higher scores indicates a worse outcome.
Changes in Life satisfaction | Change from baseline in Life Satisfaction Questionnaire to the end of the rehab program (average four month)
  Changes in Life Satisfaction measured with Life Satisfaction Questionnaire (Li-Sat-11). Minimum score at 11 and maximum score at 66. Higher scores indicate a greater level of perceived satisfaction.
Changes in Life satisfaction | Change from baseline in Life Satisfaction Questionnaire through study completion (average 1,5 years)
  Changes in Life Satisfaction measured with Life Satisfaction Questionnaire (Li-Sat-11). Minimum score at 11 and maximum score at 66. Higher scores indicate a greater level of perceived satisfaction.
Changes in Work ability | Change from baseline in Work ability to the end of the rehab program (average four month)
  Changes in work ability measured with the 7:th question in Work Ability Index questionnaire
Changes in Work ability | Change from baseline in Work ability through study completion (average 1,5 years)
  Changes in work ability measured with the 7:th question in Work Ability Index questionnaire
Changes in health-related quality of life | Change from baseline in RAND-36 to the end of the rehab program (average four month)
  Changes in health-related quality of life measured with RAND-36. The RAND-36 consists of 36 items grouped into eight multi-item scales: physical functioning (PF), role-functioning/physical (RP), pain (P), general health (GH), energy/fatigue (EF), social functioning (SF), role-functioning/emotional (RE), and emotional well-being (EW). An additional item asks about health change (HC) in the past year. Scale scores are summed and transformed into scales ranging from 0 (worst possible health state) to 100 (best possible state).
Changes in health-related quality of life | Change from baseline in RAND-36 through study completion (average 1,5 years)
  Changes in health-related quality of life measured with RAND-36. The RAND-36 consists of 36 items grouped into eight multi-item scales: physical functioning (PF), role-functioning/physical (RP), pain (P), general health (GH), energy/fatigue (EF), social functioning (SF), role-functioning/emotional (RE), and emotional well-being (EW). An additional item asks about health change (HC) in the past year. Scale scores are summed and transformed into scales ranging from 0 (worst possible health state) to 100 (best possible state).

CONTACTS AND LOCATIONS:
Overall Officials: Therese Hellman, PhD, Principal Investigator — Uppsala University
Locations (1):
- Katarina Danielsson, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No